CLINICAL TRIAL: NCT00397969
Title: Improving Surveillance for Colorectal Polyps
Brief Title: Improving the Frequency of Colonoscopy in Patients With a Previous Colorectal Polyp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard Medical School (HMS and HSDM) (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized
Other Study IDs: CDR0000492752; HMS-M11837-103; BWH-2005-P-000371/3; HPHC-1705
Record Dates: First submitted 2006-11-09; First posted 2006-11-10 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2006-12

CONDITIONS: Colorectal Cancer; Precancerous Condition
Keywords: colon cancer; rectal cancer; precancerous condition
MeSH Terms: conditions — Colorectal Neoplasms; Precancerous Conditions; Colonic Neoplasms; Rectal Neoplasms | interventions — Counseling

INTERVENTIONS:
Other: counseling intervention
Procedure: screening colonoscopy

SUMMARY:
RATIONALE: Receiving a reminder letter from their doctor may increase the frequency of colonoscopy in patients who have had a colorectal polyp removed.

PURPOSE: This randomized clinical trial is studying how well a reminder letter from their doctor improves the frequency of colonoscopy in patients who have had a colorectal polyp removed.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether rates of surveillance colonoscopy can be substantially increased by linking computerized data on endoscopic screening procedures to computerized pathology data to identify patients with prior adenomatous polyps who are due for repeat colonoscopy.
* Evaluate whether the impact of the intervention varies by patient characteristics, including age, sex, or site of primary care.

OUTLINE: This is a randomized, controlled, crossover study. Patients are stratified according to age (≤ 65 years of age vs > 65 years of age), gender, time elapsed since last colonoscopy, and primary care physician's (PCP) membership in Harvard Vanguard Medical Associates (yes vs no). Patients are randomized to 1 of 2 arms.

* Arm I: PCPs are mailed response forms (regarding the disposition of their eligible patients [e.g. patient letter mailed, patient called, scheduled for colonoscopy, colonoscopy completed elsewhere, patient refused procedure, clinical contraindication, patient deceased]) and letters reminding them that their patients are due for a follow-up colonoscopy. PCPs who do not return response forms within 4 weeks are sent a second set of reminders and patient letters.
* Arm II: Six months after the beginning of the study, PCPs are mailed response forms and patient letters once. A second set of reminders and patient letters are not sent.

PROJECTED ACCRUAL: A total of 800 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Prior diagnosis of adenomatous polyp
* Underwent prior colonoscopy with polypectomy at Brigham and Women's Hospital

  * Due for repeat colonoscopy according to current national guidelines of the American Gastroenterology Association (no colonoscopy within the past 5 years)

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2005-02; Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Successful completion of follow-up colonoscopy
Number of patients completing colonoscopy during the study period

CONTACTS AND LOCATIONS:
Overall Officials: John Ayanian, MD, MPP, Study Chair — Harvard Medical School (HMS and HSDM)
Locations (2):
- United States (2):
  - Dana-Farber/Brigham and Women's Cancer Center, Boston, Massachusetts
  - Harvard Medical School, Boston, Massachusetts

REFERENCES:
- [Derived] Ayanian JZ, Sequist TD, Zaslavsky AM, Johannes RS. Physician reminders to promote surveillance colonoscopy for colorectal adenomas: a randomized controlled trial. J Gen Intern Med. 2008 Jun;23(6):762-7. doi: 10.1007/s11606-008-0576-2. Epub 2008 Apr 2. PMID 18386103